CLINICAL TRIAL: NCT01721915
Title: A Randomized, Double-Blind, Placebo Controlled Trial to Evaluate the Effects of Vitamin D Supplementation on Metabolic and Fertility Parameters in PCOS Women
Brief Title: Vitamin D Treatment, Pharmacogenetics and Glucose Metabolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Austrian Science Fund (FWF) (Other)
Responsible Party: Principal Investigator, Lerchbaum Elisabeth, MD, A randomized, double-blind, placebo controlled trial to evaluate the effects of vitamin D, Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VitDPCOS1.0; KLI 274 (Other Grant/Funding Number: Austrian Science Fund (FWF))
Record Dates: First submitted 2012-10-31; First posted 2012-11-06 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Polycystic Ovary Syndrome; Healthy; Vitamin D Deficiency
Keywords: Polycystic Ovary Syndrome (PCOS); glucose metabolism; Vitamin D deficiency; vitamin D supplementation; pharmakogenetics; women
MeSH Terms: conditions — Polycystic Ovary Syndrome; Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D supplementation (Experimental): The treatment group will receive an oral dose of 20,000 IU vitD weekly (equivalent to 2857 IU/day) as oily drops (Oleovit D3-drops; producer: Fresenius Kabi Austria GmbH, Linz)
  Interventions: Drug: Vitamin D supplementation
- Placebo (Placebo Comparator): the placebo group will receive oily drops without vitD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D supplementation — The treatment group will receive an oral dose of 20,000 IU vitD weekly (equivalent to 2857 IU/day) as oily drops (Oleovit D3-drops; producer: Fresenius Kabi Austria GmbH, Linz)
  Other Names: A11CC05 Colecalciferol
  Arms: Vitamin D supplementation
Drug: Placebo
  Arms: Placebo

SUMMARY:
Background: Polycystic ovary syndrome (PCOS) is as common as 5-10% of all women in Austria. PCOS women frequently present with metabolic disturbances, hyperandrogenism and infertility. New therapy concepts are warranted. In our recent pilot study, vitamin D (vitD) supplementation significantly improved glucose metabolism and fertility. However, the efficacy of vitD administration shows individual variability indicating endogenous influences on pharmacological effects.

A recent genome-wide association study reported three loci (DHCR7, CYP2R1, and GC) associated with vitD insufficiency. Moreover, vitD receptor (VDR) gene variants have already been known to be associated with insulin resistance.

Aim: To test the hypothesis that vitD is efficient in changing metabolic parameters in PCOS and non-PCOS women longitudinally and to generate data on pharmacogenetic effects of vitD related genetic determinants adjusted for environmental factors.

Primary outcome: Change from baseline in AUCgluc after vitD treatment. Secondary outcome: To generate the hypothesis that changes in metabolic and endocrine parameters following vitD treatment are associated with vitD related gene variants.

Methods: 150 PCOS women with 25-hydroxyvitamin D (cholecalciferol, [25(OH)D]) levels <30 ng/ml will be treated with vitD (20,000 IU/wk) or placebo in a 2:1 randomized controlled trial over 24 weeks and investigated for metabolic and endocrine parameters as well as vitD related genetic variants. In addition, 150 non-PCOS women with 25(OH)D <30 ng/ml will be treated with vitD (20,000 IU/wk) or placebo in a 2:1 randomized controlled trial over 24 weeks and investigated for metabolic and endocrine parameters as well as vitD related genetic variants. The response to vitD supplementation in both groups will be analysed according to genotype profiles.

Significance: VitD might be a new therapeutic option without major side effects for PCOS patients. Exploring specific loci for pharmacogenetic vitD actions would open a new window for therapy modulation in PCOS and other metabolic diseases.

ELIGIBILITY:
Inclusion Criteria:

PCOS women:

* 25(OH)D levels below 30 ng/ml (measured at the baseline visit)
* Polycystic ovary syndrome defined by the Androgen Excess Society (AES) criteria
* Female, age of ≥ 18 and <45 years
* BMI status: 75 PCOS women with BMI ≤25 kg/m² and 75 PCOS women with BMI>25 kg/m²
* Written informed consent before study entry

Control women:

* 25(OH)D levels below 30 ng/ml (measured at the baseline visit)
* Female, age of ≥ 18 and <45 years
* BMI status: 75 nonPCOS women with BMI ≤25 kg/m² and 75 nonPCOS women with BMI>25 kg/m²
* Written informed consent before study entry

Exclusion Criteria:

PCOS women:

* Hypercalcemia defined as a serum calcium > 2,7 mmol/L
* Pregnancy or lactating women
* Disorders associated with androgen excess and/or menstrual irregularities apart from PCOS (thyroid dysfunction, hyperprolactinemia, adrenal hyperplasia, androgen secreting tumors)
* Prevalent type 2 diabetes
* Regular intake of vitD supplements at any time before study entry
* Intake of medication influencing metabolic or endocrine parameters (insulin sensitizers, oral contraceptives, …) in the last 3 months before study entry

Control women:

* Hypercalcemia defined as a serum calcium > 2,7 mmol/L
* Established PCOS or any of the AES criteria 29 (hyperandrogenism (clinical and/or biochemical), oligo- or anovulation, or polycystic ovaries on ultrasound)
* Disorders associated with androgen excess and/or menstrual irregularities apart from PCOS (thyroid dysfunction, hyperprolactinemia, adrenal hyperplasia, androgen secreting tumors)
* Prevalent type 2 diabetes
* Pregnancy or lactating women
* Regular intake of vitD supplements at any time before study entry
* Intake of medication influencing metabolic or endocrine parameters (insulin sensitizers, oral contraceptives, …) in the last 3 months before study entry

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 330 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2017-10-12 (Actual); Study Completion 2017-10-12 (Actual)

PRIMARY OUTCOMES:
Metabolic response during an oral glucose tolerance test (oGTT) as defined by AUCgluc | Change from Baseline in AUC gluc at 24 weeks

SECONDARY OUTCOMES:
Insulin resistance assessed by homeostatic model assessment-insulin resistance (HOMA-IR) | Change from Baseline in insulin resistance at 24 weeks
Lipid levels (total cholesterol) | Change from Baseline in total cholesterol at 24 weeks
HbA1c | Change from Baseline in HbA1c at 24 weeks
Testosterone | Change from Baseline in testosterone at 24 weeks
Menstrual frequency | Change from Baseline in menstrual frequency at 24 weeks
Insulin sensitivity assessed by Quantitative Insulin-sensitivity Check Index (QUICKI) | Change from baseline in QUICKI at 24 weeks
Free testosterone (FT) | Change from Baseline in FT at 4 weeks
Triglycerides | Change from Baseline in triglycerides at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Lerchbaum, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Department of Internal Medicine, Division of Endocrinology and Metabolism, Graz, Austria